CLINICAL TRIAL: NCT01541956
Title: An Open-labeled, Randomized, Multicenter, Prospective, Parallel Group, Interventional Study to Demonstrate the Effectiveness of 24 Weeks Treatment With Vildagliptin 50mg Bid as Add on to Metformin 500 mg Bid Compared to Metformin up to 1000 mg Bid in Chinese Patients With Type 2 Diabetes Inadequately Controlled on Metformin 500 mg Bid Monotherapy .
Brief Title: Efficacy of VIldagliptin aS an Add-on Therapy to Metformin Compared to Metformin Up-TitratION in Chinese Patients With Type 2 Diabetes.(VISION)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ACN01
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes;; vildagliptin;; metformin;
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metformin up titration (Active Comparator): metformin 500 mg bid will be up titrated (total daily dose up to 2000 mg)
  Interventions: Drug: Metformin
- vildagliptin add on to metformin (Experimental): Vildagliptin 50 mg twice daily + Metformin 500mg twice daily
  Interventions: Drug: Metformin; Drug: vildagliptin

INTERVENTIONS:
Drug: Metformin — 500 mg twice daily
Drug: vildagliptin — Vildagliptin 50 mg twice daily
  Other Names: LAF237
  Arms: vildagliptin add on to metformin

SUMMARY:
This is an open-labeled, randomized, multicenter, prospective, parallel group, interventional study to demonstrate the effectiveness of 24 weeks treatment with Vildagliptin 50mg bid as add on to metformin 500 mg bid compared to metformin up to 1000 mg bid in Chinese patients with type 2 diabetes inadequately controlled on sub maximal dosage metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Chinese T2D patients who are inadequate controlled (6.5 %< HbA1C ≤9%) by metformin (≥750mg/d but ≤1000mg/d, ≥12 weeks),

Exclusion Criteria:

* Type 1 diabetes and secondary diabetes
* Acute metabolic diabetic complications within the past 3 months.
* Acute infections which may influence glucose level.
* Evidence of significant chronic diabetic complications,
* Clinically significant renal impairment and hepatic impairment patients, including history of cirrhosis or chronic hepatitis,
* FPG > 270 mg/dl (15 mmol/l)
* Any of the following disease within the past 6 months: myocardial infarction (MI); coronary artery bypass surgery or percutaneous coronary intervention; unstable angina or stroke; Congestive heart failure (CHF)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3091 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin A1c(HbA1C) after 24 weeks of treatment with vildagliptin | baseline, 24 weeks
  The change from baseline in hemoglobin A1c(HbA1c) after 24 weeks treatment in vildagliptin 50 mg bid used in combination with metformin 500 mg bid is not inferior to that with metformin up to 1000 mg bid as monotherapy after 24 weeks

SECONDARY OUTCOMES:
Change from baseline in hemoglobin A1c(HbA1C) after 24 weeks of treatment in pre-defined patient subgroups | baseline and 24 weeks
  The changes from baseline in hemoglobin A1c(HbA1C) after 24 weeks of treatment will be analyzed in pre-defined patient subgroups based on Body Mass Index(BMI) ( <24, ≥ 24) and age (<60 y and ≥ 60 y)
Percentage of patients achieving target hemoglobin A1c( HbA1C) of ≤6.5% | baseline and 24 weeks
  The percentage of patients achieving target hemoglobin A1c( HbA1C) of ≤6.5% of two treatment arms in the overall population and in pre defined sub groups.
Percentage of patients achieving target hemoglobin A1c(HbA1C) of ≤6.5% without adverse gastrointestinal (GI) events | baseline and 24 weeks
  The percentage of patients achieving target hemoglobin A1c( HbA1C) of ≤6.5% without adverse GI events of two treatment arms in the overall population and in pre defined sub groups.
Mean change from baseline in fasting plasma glucose (FPG) | baseline, 24 weeks
  Mean change from baseline in FPG will be calculated in the overall population and in pre defined sub groups.
Mean change from baseline in 2-hour post prandial glucose( PPG) in a sub sample | baseline, 24 weeks
  Mean change from baseline in 2 hour post prandial glucose(PPG) in a sub sample of overall patients.
Number of patients with adverse events, serious adverse events and death | up to 24 weeks
  Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Beijing, China

REFERENCES:
- [Result] Ji LN, Pan CY, Lu JM, Li H, Zhu DL, Li Q, Li QF, Peng YD, Tian HM, Yao C, Zhao ZG, Wang L, Wang BH; VISION Study Group. Efficacy and safety of combination therapy with vildagliptin and metformin versus metformin uptitration in Chinese patients with type 2 diabetes inadequately controlled with metformin monotherapy: a randomized, open-label, prospective study (VISION). Diabetes Obes Metab. 2016 Aug;18(8):775-82. doi: 10.1111/dom.12667. Epub 2016 May 18. PMID 27406394